CLINICAL TRIAL: NCT03522454
Title: Protein and Exercise to Reverse Frailty in OlderR Men and Women Undergoing TAVR: The PERFORM-TAVR Trial
Brief Title: The PERFORM-TAVR Trial
Acronym: PERFORM-TAVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: University of British Columbia (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); St. Boniface Hospital (Other); Montreal Heart Institute (Other); Hamilton Health Sciences Corporation (Other); Ottawa Heart Institute Research Corporation (Other); Unity Health Toronto (Other); Sunnybrook Research Institute (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Jonathan Afilalo, Principal Investigator, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 378469
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Frail Elderly; Exercise; Dietary Supplements; Postoperative Care; Rehabilitation; Transcatheter Aortic Valve Replacement
Keywords: Frailty; TAVR
MeSH Terms: conditions — Motor Activity; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor who will perform the 3 and 6 month visits will be blinded to the participant's assigned intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: Combination of a protein-rich oral nutritional supplement consumed twice daily for 4 weeks pre-TAVR and 12 weeks after the patient is discharged home post-TAVR, and a home-based supervised exercise program that combines walking and weight-bearing exercises to build strength and balance performed for 12 weeks after the patient is discharged home post-TAVR.
  Interventions: Dietary Supplement: Protein-rich oral nutritional supplement; Behavioral: Home-based supervised exercise program
- Lifestyle counselling group (No Intervention): Lifestyle counselling group: Recommendation to perform moderate-intensity aerobic activity at least 30 minutes 5 days per week as tolerated and eat a balanced diet based on the AHA/ACC Guideline on Lifestyle Management.

INTERVENTIONS:
Dietary Supplement: Protein-rich oral nutritional supplement — Ready-to-drink beverage containing 20 g protein and 1.5 g hydroxymethylbutyrate (HMB) per serving, consumed twice daily.
  Arms: Intervention group
Behavioral: Home-based supervised exercise program — WEBB (Weight-bearing Exercise for Better Balance) program combining walking and weight-bearing exercises to build strength and balance, administered by a trained therapist at the participant's home.
  Arms: Intervention group

SUMMARY:
The PERFORM-TAVR trial (Protein and Exercise to Reverse Frailty in OldeR Men and women undergoing Transcatheter Aortic Valve Replacement) is a multicenter randomized clinical trial with a parallel-group design. The investigators will screen consecutive patients ≥70 years of age before TAVR and enrol those that have evidence of physical frailty defined by an SPPB score ≤8 or an SF36-PF score ≤55. The investigators will randomly allocate 200 patients to receive a multi-faceted intervention consisting of a home-based exercise program and a protein-rich oral nutritional supplement or usual lifestyle counselling. The primary endpoint will be the change in SF36-PF score at 12 weeks.

DETAILED DESCRIPTION:
STUDY DESIGN:

The PERFORM-TAVR trial (Protein and Exercise to Reverse Frailty in OldeR men and woMen undergoing Transcatheter Aortic Valve Replacement) is a multicenter randomized clinical trial with a parallel-group design. We will screen consecutive patients ≥70 years of age before TAVR and enroll those that have evidence of physical frailty defined as an SPPB score ≤8 or an SF36-PF score ≤55. The SPPB and SF36-PF were chosen as the main inclusion criteria and also as key endpoints based on their ease-of-use, reproducibility, responsiveness to change, and superior predictive value for mortality and patient-centered outcomes in the Frailty-AVR Study. We will randomly allocate 200 patients to receive a multi-faceted intervention consisting of home-based exercise and protein supplementation or standard-of-care lifestyle counselling.

INTERVENTION GROUP:

The multi-faceted intervention consists of two synergistic components performed by participants at their homes. The first component is a home-based supervised exercise program that combines walking and weight-bearing exercises to build strength and balance performed for 12 weeks after the patient is discharged home post-TAVR. The exercises are based on the WEBB program that was developed at the University of Sydney and validated to help therapists individually prescribe progressive exercise that is challenging but safe for older adults (http://www.webb.org.au/attachments/File/WEBB_draft_19.pdf). Starting as soon as the patient returns home post-TAVR, a trained therapist (TT; physiotherapist or certified exercise physiologist, depending on local expertise) will visit their home for 1 hour twice weekly over a 12-week period to supervise and tailor the exercises according to each individual's capability and progress, and to reinforce the goal of moderate-intensity aerobic activity such as brisk walking at least 30 minutes 5 days per week. If the patient is transferred to a convalescence or inpatient rehabilitation facility or another hospital, the TT will defer home visits until they are discharged to their home. If the patient is referred to an outpatient rehabilitation program, the TT will continue to perform home visits concurrently. The low use of center-based rehabilitation reflects well-known accessibility barriers in our Canadian healthcare environment and reaffirms the high relevance of our home-based intervention.

To monitor compliance, the TT will ask patients to note their daily exercises in their log book and wear a wrist-worn accelerometer (Garmin Vivofit 4) to record daily step counts. The accelerometer provides motivational cues such as individualized daily step count goals and gentle beeps to remind patients to move when they have been sedentary for a prolonged period during the day. We previously used the Garmin Vivofit in an elderly cardiac population as part of the Get Going Trial and found it to be "geriatric-friendly" owing to its minimalist interface, large font size, lightweight waterproof design, and year-long battery that does not necessitate charging or computer syncing. The majority of patients (including those ≥80 years) reported a high level of comprehension and satisfaction with this device. The TT will sync the patient's accelerometer devices at every home visit using a smartphone or tablet, review their step counts, and provide personalized coaching to increase daily walking.

The second component is a protein-rich oral nutritional supplement (Ensure Enlive) with 20g protein and 1.5g HMB per serving, delivered as a ready-to-drink beverage in 235 mL bottles, consumed twice daily for 4 weeks pre-TAVR and 12 weeks after the patient is discharged home post-TAVR. This beverage contains 350 calories, and is provided in chocolate and vanilla flavors. It should be consumed with breakfast (first serving of the day) and with exercise (second serving of the day), not before meals, so as to supplement rather than replace food intake. The HMB ingredient stimulates muscle protein synthesis, particularly when combined with exercise due to the muscle priming effect. To monitor and promote compliance, the TT will ask patients to note their beverage consumption in their log book, instruct them to consume a beverage during home exercise sessions, periodically replenish their supply of beverages during home visits, and perform bottle counts. The log book provided to the participants also contains information on healthy eating and maintaining an active lifestyle (same as control group).

LIFESTYLE COUNSELLING GROUP:

Lifestyle counselling consists of formalized usual care - instructing patients to perform moderate-intensity aerobic activity at least 30 minutes 5 days per week as tolerated and eat a balanced diet based on the AHA/ACC Guideline on Lifestyle Management. In order to standardize this counselling and ensure that it is safely carried out in both groups, the TT will provide and explain information on healthy eating and maintaining an active lifestyle based on the "Easy Tips for Heart Healthy Eating" and "Walking for a Healthy Heart" brochures designed by the American Heart Association. The latter outlines practical tips to safely begin a walking program and gradually increase walking time over a 12-week period to meet the goal of 150 minutes per week. All of this information will be easily legible in a log book provided to participants. We will not instruct lifestyle counselling group patients to consume protein-rich nutritional supplements during the trial unless prescribed by their treating physician.

OUTCOME MEASURES:

The primary endpoint is the SF36-PF score at 12 weeks. Secondary endpoints are physical functioning measured by the Short Physical Performance Battery (SPPB), health-related QOL measured by the 36-Item Short Form Health Survey (SF-36), cognitive function measured by the Montreal Cognitive Assessment (MoCA), habitual physical activity level measured by the modified Paffenbarger questionnaire, handgrip strength measured by a Jamar dynamometer, body composition and phase angle measured by a portable bioimpedance device, frailty measured by the Essential Frailty Toolset, sarcopenia measured by the SARC-F questionnaire and EWGSOP criteria, and a composite safety endpoint of all-cause mortality, injurious fall, acute kidney injury, or readmission for worsening angina, heart failure, or arrhythmia. The aforementioned primary and secondary endpoints will be re-assessed at 24 weeks to detect latent effects and sustained adherence, and vital status and questionnaires will be assessed by telephone at 52 weeks. Clinical events will be defined according to the Valve Academic Research Consortium-2 data dictionary. A 3-member independent Data Safety and Monitoring Board will review all adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Undergoing TAVR
* Physically frail: SPPB score ≤8 or SF36-PF score ≤ 55 pre-TAVR
* Informed written or verbal consent

Exclusion Criteria:

* Decompensated or non-ambulatory class IV symptoms of angina, dyspnea, claudication
* Uncontrolled diabetes with HbA1C >8.5% (or mean glucose ≥11.0 in the absence of a HbA1C test)
* Glomerular filtration rate (GFR) <30 mL/min/1.73 m2 by the MDRD equation
* Cirrhosis
* Allergy to ingredient in beverage
* Inability to safely ingest beverage by mouth
* Inability to walk without human assistance or high-risk of falls
* Moderate-to-severe cognitive impairment
* Significant language barrier
* COVID positive or suspected at screening

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
SF36-PF | 3 months
  Short-Form 36 Physical Functioning (SF36-PF) scale; range 0-100 (higher is better)

SECONDARY OUTCOMES:
SPPB | 3 and 6 months
  Short Physical Performance Battery (SPPB) scale; range 0-12 (higher is better)
Health-related quality of life | 3, 6, and 12 months
  Short Form Health Survey (SF-36) scale; population-standardized to mean score of 50 with standard deviation of 10 (higher is better) for the 8 section scores and 2 summary scores
Habitual physical activity (in kcal per week) | 3, 6, and 12 months
  Modified Paffenbarger activity scale; range 0-upwards (higher is better)
Frailty | 3 and 6 months
  Essential Frailty Toolset (EFT) scale; range 0-5 (lower is better)
Sarcopenia | 3, 6, and 12 months
  SARC-F scale; range 0-10 (lower is better)
Fat free mass (in kg) | 3 and 6 months
  Portable bioimpedance device; biological range (higher is better)
Phase angle (in degrees) | 3 and 6 months
  Portable bioimpedance device; biological range (higher is better)
Handgrip strength (in kg) | 3 and 6 months
  Jamar dynamometer; range 0-upwards (higher is better)
Cognitive function | 3 and 6 months
  Montreal Cognitive Assessment (MoCA) scale; range 0-30 (higher is better)
Number of participants suffering composite safety endpoint | 3 and 6 months
  All-cause mortality, injurious fall, acute kidney injury, or readmission for worsening angina, heart failure, or arrhythmia
Number of participants suffering death from any cause | 3, 6, and 12 months
  All-cause mortality assessed by medical records and telephone contact

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Afilalo, MD, MSc, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital / McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fountotos R, Lauck S, Piazza N, Martucci G, Arora R, Asgar A, Forcillo J, Kouz R, Labinaz M, Lamy A, Peterson M, Wijeysundera H, Masse L, Ouimet MC, Polderman J, Webb J, Afilalo J. Protein and Exercise to Reverse Frailty in Older Men and Women Undergoing Transcatheter Aortic Valve Replacement: Design of the PERFORM-TAVR Trial. Can J Cardiol. 2024 Feb;40(2):267-274. doi: 10.1016/j.cjca.2023.11.037. Epub 2023 Dec 3. PMID 38052302